CLINICAL TRIAL: NCT07208747
Title: Construction and Application of an Intelligent Module for Pressure Injury Nursing Management System
Brief Title: Evaluating an Intelligent Module for Pressure Injury Nursing Management
Acronym: IM-PINM
Status: Completed | Type: Observational
Sponsor: Xiamen Humanity Hospital (Other)
Responsible Party: Principal Investigator, CHAO JING, Deputy Chief Nurse, Xiamen Humanity Hospital
Other Study IDs: HAXM-MEC-20250815-069-01
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Pressure Injury
Keywords: Pressure injury；Nursing management system；Intelligent module
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed Cohort: The nursing staff routinely used the intelligent pressure-injury management module as part of standard care throughout 2024.
- Routine Care Cohort: The nursing staff provided routine pressure-injury care without the use of the intelligent module throughout 2023.

SUMMARY:
This is a study conducted in a hospital to evaluate whether applying an intelligent information technology can help nurses better prevent and manage bedsores (also known as pressure injuries) in hospitalized patients. Bedsores are a serious skin problem for patients who are bedridden for long periods. The researchers will compare the situation before and after using the intelligent program to see if it has an impact on the occurrence and outcomes of pressure injuries. We invite eligible hospitalized patients to participate. Participants' nursing data will be anonymously recorded and analyzed to evaluate the effectiveness of this intelligent program.

DETAILED DESCRIPTION:
Background：Pressure injuries are common nursing complications in clinical practice, and their occurrence can reduce patients' quality of life, affect rehabilitation, and increase medical costs. This project aims to utilize information technology to build a comprehensive and intelligent pressure injury care management platform, providing scientific evidence for clinical decision-making and supporting standardized management of pressure injuries and improvement in nursing quality.

Objective：To construct an intelligent module for the pressure injury nursing management system and to explore its application effects in pressure injury management.

Methods：Based on the hospital nursing information system, an intelligent module was constructed to achieve functions such as intelligent decision-making for pressure injury risk assessment, intelligent staging judgment, visual online assessment and review, outcome tracking，and home care linkage, as well as monitoring quality control indicators.

ELIGIBILITY:
Inclusion Criteria:

* Length of stay ≥ 2 hours after admission

Exclusion Criteria:

* 1: Terminal condition (expected survival time < 48 hours) 2: Refusal to participate in data collection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients admitted to the Xiamen Humanity Hospital during 2023 and 2024.
Sampling Method: Non-Probability Sample
Enrollment: 75263 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Braden scale assessment timeliness rate(≤2hours from admission) | The time frame for data collection is from January 2023 to December 2024, with data collected monthly.
  1.Number of newly admitted patients assessed within 2 h: The system automatically pulls timestamps from the Nursing Management System-start time = patient's arrival timestamp; end time = nurse's submission timestamp of the Braden assessment. Records with an interval ≤ 2 h are counted as "timely." 2.Total newly admitted patients in the period: The system extracts the total number of patients who completed admission procedures. 3.Formula:Braden Risk Assessment Timeliness Rate = (number of newly admitted patients assessed within 2 h ÷ total newly admitted patients in the period) × 100%
Braden Assessment omission rate | The time frame for data collection is from January 2023 to December 2024, with data collected monthly.
  1.The required assessments based on the patient's Braden score: ≥19 (no risk): once on admission and once on discharge 15-18 (low risk): once per week 13-14 (moderate risk): twice per week (re-assessed on Tuesday and Friday) 10-12 (high risk): once per day 0-9 (very high risk): once per nursing shift (three shifts) Actual assessments: The assessments recorded in the nursing system. Missed assessments= required assessments - actual assessments 2.Formula:Braden Assessment Omission Rate =Missed assessments (required count - actual count) ÷ Required count
Accuracy rate in PI staging determination | The time frame for data collection is from January 2023 to December 2024, with data collected monthly.
  1.The system automatically pulls from the Nursing Management Information System all in-hospital and community-acquired pressure injury (PI) reports submitted every month. The wound-care specialists then identify-per NPUAP/EPUAP staging criteria-those records whose initial stage was judged "incorrect." 2.Total Reports: The system simultaneously extracts the total number of all PI reports submitted during the same month. 3.Formula: PI staging accuracy (%) = (correctly staged cases ÷ total reported cases) × 100%.

SECONDARY OUTCOMES:
Hospital-Acquired Pressure Injury (HAPI) Incidence Rate | The time frame for data collection is from January 2023 to December 2024, with data collected monthly.
  1."Monthly incident cases": Automatically extracted each month from the Nursing Management System-counts all newly acquired pressure injuries that have been reported during the month. "Total inpatient episodes for the same period": Simultaneously extracted the total cumulative inpatient episodes for the month, including transfers and deaths; same-day readmissions are counted only once. 3.Formula: Hospital-acquired pressure injury incidence (%) = (monthly new hospital-acquired cases ÷ monthly total inpatient episodes) × 100%.
Wound outcome classification | The time frame for data collection is from January 2023 to December 2024, with data collected annually.
  1. Annual wound outcome records: The system automatically pulls the wound outcome fields (healed / improved / unchanged / deteriorated) for all discharged patients with PIs in per year. 2.Total number of PI patients: The sum of all hospital-acquired plus community-acquired pressure injury cases in the same year, denoted as N. 3.Formula: • Healing rate (%) = (number of healed cases ÷ N) × 100% Improvement rate (%) = (number of improved cases ÷ N) × 100% Unchanged rate (%) = (number of unchanged cases ÷ N) × 100% Deterioration rate (%) = (number of deteriorated cases ÷ N) × 100%

CONTACTS AND LOCATIONS:
Locations (1):
- Xiamen Humanity Hospital, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
1. De-identified individual participant data that underlie the results reported in this article will be shared after the publication of the primary findings.
  2. Researchers who provide a methodologically sound proposal will be granted access. Proposals should be directed to water1427@sina.com. To gain access, requestors will need to sign a data access agreement.
  3. The data will be made available for at least 5 years. We aim to provide data within 5 business days of request approval.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting documents will become available after the publication of the primary results manuscript for a period of at least 5 years.
Access Criteria: Data will be available to researchers who provide a scientifically sound research proposal that has been approved by an independent review committee. Proposals should be directed to the corresponding author (water1427@sina.com). Access will be granted after the signing of a data access agreement that includes commitments to: 1) use the data only for the specified research purpose; 2) not attempt to re-identify participants; 3) secure the data appropriately.